CLINICAL TRIAL: NCT02293551
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Novel Insulin Lispro Formulations
Brief Title: A Study of Lispro Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15626; F3Z-FW-ITCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A: Lispro (A) (Experimental): Formulation A: Single dose of lispro administered subcutaneously (SC) in one of five periods.
  Interventions: Drug: Lispro
- Part A: Lispro (B) (Experimental): Formulation B: Single dose of lispro administered SC in one of five periods.
  Interventions: Drug: Lispro
- Part A: Lispro (C) (Experimental): Formulation C: Single dose of lispro administered SC in one of five periods.
  Interventions: Drug: Lispro
- Part A: Lispro (D) (Experimental): Formulation D: Single dose of lispro administered SC in one of five periods.
  Interventions: Drug: Lispro
- Part A: Lispro (Reference) (Experimental): Reference formulation: Single dose of lispro administered SC in one of five periods.
  Interventions: Drug: Lispro
- Part B: Lispro (Experimental): Formulation selected from Part A. Single dose of lispro administered SC in one of four periods.
  Interventions: Drug: Lispro

INTERVENTIONS:
Drug: Lispro — Administered SC
  Other Names: LY275585

SUMMARY:
The purposes of this study are to determine:

* Part A

  * How quickly your body absorbs, breaks down and gets rid of the different formulations of insulin lispro compared to insulin lispro alone formulation.
  * The safety of insulin lispro in different formulations and any side effects that might be associated with it.
* Part B:

  * How much insulin lispro from different dose ranges is found in the bloodstream using a test insulin lispro formulation (selected from Part A).
  * The safety of insulin lispro in different formulations and any side effects that might be associated with it.

Participants may only enroll in one part. The study is expected to last up to 10 weeks for each part.

ELIGIBILITY:
Inclusion Criteria:

- Overtly healthy males or females (non-childbearing potential and with absent cyclical hormonal changes), as determined by medical history and physical examination

Exclusion Criteria:

- Have a fasting plasma glucose less than or equal to (≤) 4.0 millimole per liter (mmol/L) at screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A was a 5-period crossover study and Part B was a 4-period crossover study. A washout of 72 hours was observed between doses with a follow up within 7 to 14 days after the last dose.
Groups:
- Part A: Lispro Sequence 1: Each participant received a single subcutaneous (SC) dose of 7.0 U insulin lispro (Reference) and 4 doses of different test insulin lispro formulations (7.28 U; Tests A, B, C, and D) in one of five periods according to assigned treatment sequence 1, 2, or 3.
  Sequence 1: Test A, D, C, Reference, B
- Part A: Lispro Sequence 2: Each participant received a single SC dose of 7.0 U insulin lispro (Reference) and 4 doses of different test insulin lispro formulations (7.28 U; Tests A, B, C, and D) in one of five periods according to assigned treatment sequence 1, 2, or 3.
  Sequence 2: Test B, A, Reference, C, D
- Part A: Lispro Sequence 3: Each participant received a single SC dose of 7.0 U insulin lispro (Reference) and 4 doses of different test insulin lispro formulations (7.28 U; Tests A, B, C, and D) in one of five periods according to assigned treatment sequence 1, 2, or 3.
  Sequence 3: Test Reference, Test C, B, D, A.
- Part B: Lispro Sequence 1: Each participant received a single dose of lispro SC in one of four periods according to assigned treatment sequence 1, 2, or 3. Participants received test formulation B containing 7.28 U (Units) of insulin lispro given as a single SC injection or test formulation B containing 15.47 U of insulin lispro given as a single SC injection or test formulation B containing 30.03 U of insulin lispro given as a single SC injection.
  Sequence 1: 30.03 U, 7.28 U, 15.47 U, 7.28 U
- Part B Lispro Sequence 2: Each participant received a single dose of lispro SC in one of four periods according to assigned treatment sequence 1, 2, or 3. Participants received test formulation B containing 7.28 U (Units) of insulin lispro given as a single SC injection or test formulation B containing 15.47 U of insulin lispro given as a single SC injection or test formulation B containing 30.03 U of insulin lispro given as a single SC injection.
  Sequence 2: 7.28 U, 15.47 U, 30.03 U, 15.47 U
- Part B Lispro Sequence 3: Each participant received a single dose of lispro SC in one of four periods according to assigned treatment sequence 1, 2, or 3. Participants received test formulation B containing 7.28 U (Units) of insulin lispro given as a single SC injection or test formulation B containing 15.47 U of insulin lispro given as a single SC injection or test formulation B containing 30.03 U of insulin lispro given as a single SC injection.
  Sequence 3: 15.47 U, 30.03 U, 7.28 U, 30.03 U
Period: Part A and Part B Period 1
Arm/Group | Part A: Lispro Sequence 1 | Part A: Lispro Sequence 2 | Part A: Lispro Sequence 3 | Part B: Lispro Sequence 1 | Part B Lispro Sequence 2 | Part B Lispro Sequence 3
Started | 8 | 8 | 8 | 10 | 10 | 10
Completed | 8 | 8 | 8 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A and B Period 2
Arm/Group | Part A: Lispro Sequence 1 | Part A: Lispro Sequence 2 | Part A: Lispro Sequence 3 | Part B: Lispro Sequence 1 | Part B Lispro Sequence 2 | Part B Lispro Sequence 3
Started | 8 | 8 | 8 | 10 | 10 | 10
Completed | 8 | 8 | 8 | 10 | 10 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Part A and B Period 3
Arm/Group | Part A: Lispro Sequence 1 | Part A: Lispro Sequence 2 | Part A: Lispro Sequence 3 | Part B: Lispro Sequence 1 | Part B Lispro Sequence 2 | Part B Lispro Sequence 3
Started | 8 | 8 | 8 | 10 | 10 | 9
Completed | 8 | 8 | 8 | 8 | 10 | 8
Not Completed | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 1
Period: Part A and Part B Period 4
Arm/Group | Part A: Lispro Sequence 1 | Part A: Lispro Sequence 2 | Part A: Lispro Sequence 3 | Part B: Lispro Sequence 1 | Part B Lispro Sequence 2 | Part B Lispro Sequence 3
Started | 8 | 8 | 8 | 8 | 10 | 8
Completed | 8 | 8 | 8 | 6 | 10 | 7
Not Completed | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 1
Period: Part A Period 5
Arm/Group | Part A: Lispro Sequence 1 | Part A: Lispro Sequence 2 | Part A: Lispro Sequence 3 | Part B: Lispro Sequence 1 | Part B Lispro Sequence 2 | Part B Lispro Sequence 3
Started | 8 | 8 | 8 | 0 (Part B had 4 periods) | 0 (Part B had 4 periods) | 0
Completed | 8 | 8 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A Participants: Each participant received a single SC dose of 7.0 U insulin lispro (Reference) and 4 doses of different test insulin lispro formulations (7.28 U; Tests A, B, C, and D) in one of five periods according to assigned treatment sequence 1, 2, or 3.
  Sequence 1: Test A, D, C, Reference, B Sequence 2: Test B, A, Reference, C, D Sequence 3: Test Reference, Test C, B, D, A.
- Part B Participants: Each participant received a single dose of lispro SC in one of four periods according to assigned treatment sequence 1, 2, or 3. Participants received test formulation B containing 7.28 U (Units) of insulin lispro given as a single SC injection or test formulation B containing 15.47 U of insulin lispro given as a single SC injection or test formulation B containing 30.03 U of insulin lispro given as a single SC injection.
  Sequence 1: 30.03 U, 7.28 U, 15.47 U, 7.28 U Sequence 2: 7.28 U, 15.47 U, 30.03 U, 15.47 U Sequence 3: 15.47 U, 30.03 U, 7.28 U, 30.03 U
- Total: Total of all reporting groups
Arm/Group | Part A Participants | Part B Participants | Total
Number analyzed (Participants) | 24 | 30 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (11.5) | 36.8 (9.1) | 37.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 30 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 30 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 27 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 3 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 24 | 30 | 54

OUTCOME MEASURES:

1. Primary Outcome: Part A and Part B: Pharmacokinetics (PK): Area Under The Concentration Curve Zero to Infinity (AUC[0-∞])
Description: Primary outcome measure is based on the PK area under the concentration curve from 0 to infinity with a measurable concentration.
Time Frame: -30, 0 (Predose), 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150,180, 240, and 300 Minutes
Population: All randomized participants who were completers and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole*hour/Liter (pmol*hr/L)
Groups:
- Part A: Lispro (7.0 U - Reference): Reference formulation: Single dose of lispro administered SC in one of five periods.
- Part A: Lispro (7.28 U - Test A): Formulation A: Single dose of lispro administered SC in one of five periods.
- Part A: Lispro (7.28 U - Test B): Formulation B: Single dose of lispro administered SC in one of five periods.
- Part A: Lispro (7.28 U - Test C): Formulation C: Single dose of lispro administered SC in one of five periods.
- Part A: Lispro (7.28 U - Test D): Formulation D: Single dose of lispro administered SC in one of five periods.
- Part B: Lispro (7.28 U - Test B); Part B: Lispro (15.47 U - Test B); Part B: Lispro (30.03 U - Test B): Formulation selected from Part A. Single dose of lispro administered SC in one of four periods.
Arm/Group | Part A: Lispro (7.0 U - Reference) | Part A: Lispro (7.28 U - Test A) | Part A: Lispro (7.28 U - Test B) | Part A: Lispro (7.28 U - Test C) | Part A: Lispro (7.28 U - Test D) | Part B: Lispro (7.28 U - Test B) | Part B: Lispro (15.47 U - Test B) | Part B: Lispro (30.03 U - Test B)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 28 | 28 | 29
picomole*hour/Liter (pmol*hr/L) | 916 (21) | 957 (22) | 1020 (22) | 972 (21) | 971 (23) | 864 (17) | 2000 (20) | 3990 (14)
Statistical Analysis 1: Comparison: Part A: Lispro (7.0 U - Reference) vs Part A: Lispro (7.28 U - Test A); Test type: Superiority or Other; p = 0.2071, Log Rank; Log (PK) model included treatment, period, and sequence group as fixed effects and participant as a random effect; Geometric Ratio of Least Squares Mean = 1.04, 90% CI 2-sided [0.988 to 1.10]
Statistical Analysis 2: Comparison: Part A: Lispro (7.0 U - Reference) vs Part A: Lispro (7.28 U - Test B); Test type: Superiority or Other; p = 0.0005, Log Rank; Log (PK) model included treatment, period, and sequence group as fixed effects and participant as a random effect; Geometric Ratio of Least Square Means = 1.11, 90% CI 2-sided [1.06 to 1.17]
Statistical Analysis 3: Comparison: Part A: Lispro (7.0 U - Reference) vs Part A: Lispro (7.28 U - Test C); Test type: Superiority or Other; p = 0.0123, Log Rank; Log (PK) model included treatment, period, and sequence group as fixed effects and participant as a random effect; Geometric of Ratio Least Square Means = 1.08, 90% CI 2-sided [1.03 to 1.13]
Statistical Analysis 4: Comparison: Part A: Lispro (7.0 U - Reference) vs Part A: Lispro (7.28 U - Test D); Test type: Superiority or Other; p = 0.0331, Log Rank; Log (PK) model included treatment, period, and sequence group as fixed effects and participant as a random effect; Geometric Ratio of Least Square Means = 1.07, 90% CI 2-sided [1.02 to 1.13]
Statistical Analysis 5: Comparison: Part B: Lispro (7.28 U - Test B) vs Part B: Lispro (15.47 U - Test B) vs Part B: Lispro (30.03 U - Test B); Test type: Superiority or Other; Mean Difference (Final Values) = 1.11, 90% CI 2-sided [1.06 to 1.16] — Dose proportionality and the degree of dose proportionality was assessed by fitting the power model versus dose. Estimated ratio of dose-normalized geometric means of PK parameters between the highest and lowest doses assessed dose proportionality

ADVERSE EVENTS:
Description: 54 participants were randomly assigned to treatment, 54 participants received at least 1 dose of study drug, 24 participants completed all 5 periods of the study.
Groups:
- Part B: Lispro (7.28 U - Test B); Part B: Lispro (15.47 U - Test B); Part B: Lispro (30.03 U - Test B): Formulation selected from Part B. Single dose of lispro administered SC in one of four periods.
Arm/Group | Part A: Lispro (7.0 U - Reference) | Part A: Lispro (7.28 U - Test A) | Part A: Lispro (7.28 U - Test B) | Part A: Lispro (7.28 U - Test C) | Part A: Lispro (7.28 U - Test D) | Part B: Lispro (7.28 U - Test B) | Part B: Lispro (15.47 U - Test B) | Part B: Lispro (30.03 U - Test B)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/28 | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 4/24 | 4/24 | 4/24 | 4/24 | 2/24 | 6/28 | 3/28 | 7/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Lispro (7.0 U - Reference) (N=24) | Part A: Lispro (7.28 U - Test A) (N=24) | Part A: Lispro (7.28 U - Test B) (N=24) | Part A: Lispro (7.28 U - Test C) (N=24) | Part A: Lispro (7.28 U - Test D) (N=24) | Part B: Lispro (7.28 U - Test B) (N=28) | Part B: Lispro (15.47 U - Test B) (N=28) | Part B: Lispro (30.03 U - Test B) (N=29)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Catheter site related reaction (General disorders) | 3 (6) | 2 (3) | 4 (4) | 2 (3) | 0 (0) | 5 (5) | 2 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No